CLINICAL TRIAL: NCT01359085
Title: Pain Relief Following Arthroscopic Rotator Cuff Repair: Perioperative Pregabalin Administration Versus Interscalene Brachial Plexus Block. a Prospective, Randomized, Double Blinded, Multicenter Trial
Brief Title: Pain Relief Following Arthroscopic Rotator Cuff Repair: Perioperative Pregabalin Administration Versus Interscalene Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Helena Farladansky, MD, Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TASMC-11-HF-0235-11-CTIL
Record Dates: First submitted 2011-05-18; First posted 2011-05-24 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Pain
Keywords: To compare postoperative pain relief by pregabalin versus ISBPB following arthroscopic rotator cuff repair; To compare postoperative opioid consumption and opioid related AEs; To compare patients recovery profile and patients satisfaction
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin
- ISBPB (Active Comparator): Interscalene brachial plexus block
  Interventions: Procedure: ISBPB - interscalene brachial plexus block

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 75 mg will be given orally as premedication at the night before surgery (at bedtime). Pregabalin 150 mg will be administered orally at 1h preoperatively and at 12h and 24h postoperatively.
  Arms: Pregabalin
Procedure: ISBPB - interscalene brachial plexus block — ISBPB will be performed by an anesthesiology consultant experienced in performing the procedure, after the induction of GA. Block will be performed under sterile conditions by injection of 40ml 0.5% bupivacaine with epinephrine 1:100,000 to the plexus sheath through a 5-cm, 23-gauge short-beveled needle.
  Arms: ISBPB

SUMMARY:
Arthroscopic rotator cuff (RC) repair is often associated with severe post operative pain and discomfort. Many analgesic protocols have been proposed for pain relief following RC repair and controversy remains regarding the optimal postoperative analgesic protocol. Despite significant advancement in analgesic techniques over the last decades 50-70% of patients who undergo surgical procedures still experience moderate to severe postoperative pain. Postoperative pain has both inflammatory component (i.e. related to traumatic tissue damage and inflammatory reaction due to the surgical incision and procedure) and neuropathic component (i.e. related to over sensitization of the peripheral and central nervous system). Opioids are commonly used for postoperative pain reduction, however their use is associated with numerous adverse events and should be limited.

Regional nerve block techniques have been emerged over the past decade and have become a standard of practice recently. Recent studies indicate that a single-dose interscalene brachial plexus block (ISBPB) is effective in providing postoperative analgesia following shoulder surgery, reduces the need for opioid medication, and has a very high success rates (≥94%) and few major complications (≤0.4%). However, regional nerve blockade, including ISBPS, has a frequent incidence of temporary postoperative neurological symptoms within the first postoperative week (4 -16%), is technically demanding and might be time consuming.

Pregabalin (Lyrica) is an anticonvulsant drug with membrane stabilizing and anti-nociceptive effects commonly used for neuropathic pain relief and anxiety disorder. It desensitizes the presynaptic terminals of hyperexcited neurons in peripheral and central nervous system (i.e. reduces the transmission of excitatory neurotransmitters including glutamate, norepinephrine, substance P, and calcitonin gene-related peptide) by reducing calcium influx through high-voltage-activated calcium channels containing the alpha2/delta subunit. Pregabalin is rapidly absorbed from the gut with bioavailability of approximately 90%, achieves peak plasma concentration approximately 1h after administration, has half-life of about 6h and is eliminated by renal excretion. Many studies over the past decade have evaluated pregabalin roll in the treatment of acute postoperative pain. Pregabalin effect in reducing opioid consumption and opioid adverse events (AEs) has been well established. Its analgesic effect on acute postoperative pain remains questionable, and further studies are still required to compare pregabalin analgesic potential with other standard post-operative analgesic regimens. Pregabalin doses used in previous studies ranged from 75 to 600 mg given as a single dose 1-2h preoperatively with or without additional doses at 12h and 24h postoperatively. Doses of 150 mg and higher seemed to offer better results in terms of postoperative analgesia and opioids sparing. However higher doses were associated with higher rate of AEs, mainly sedation, dizziness and visual disturbances.

Nervous system desensitization by oral medication (e.g. pregabalin) rather than by invasive means (e.g. ISBPB) may reduce adverse reactions, increase patient satisfaction and save valuable time in the operation theater. To the investigators knowledge no previous study has compared the efficacy of pregabalin to ISBPB for acute pain relief following arthroscopic shoulder surgery. The investigators hope to contribute to the discussion regarding the optimal pain relief method following arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III patients (> 18 years old) with normal renal and coagulation function, scheduled for elective arthroscopic RC repair at Tel Aviv-Sourasky Medical Center or Tel Aviv Assuta Medical Center shoulder surgery unit.

Exclusion Criteria:

* Patients with known pulmonary or renal disease
* Known preexisting neurological disorders involving the operative limb
* Known hypersensitivity to the medication used in the study
* Considerable tension on the repair site requiring application of an abduction splint (on the discretion of the surgeon) and pregnant women will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
To compare postoperative pain relief by pregabalin versus ISBPB following arthroscopic rotator cuff repair | 1 year
  Clinical parameters (pain, satisfaction, recovery, opioid consumption and AE) will be assessed at arriving to the recovery unit, at 12h and 24h postoperatively and in days 2 and 7 postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Weizman 6, Israel